CLINICAL TRIAL: NCT04285229
Title: A Multicenter, Randomized, Double-Blind and Placebo-Controlled 16-Week Study Followed by Long Term Evaluation of Efficacy and Safety of Ixekizumab (LY2439821) in Chinese Patients With Radiographic Axial Spondyloarthritis
Brief Title: A Study of Ixekizumab (LY2439821) in Chinese Participants With Radiographic Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16721; I1F-MC-RHCH (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Spondyloarthritis
Keywords: Ankylosing spondylitis
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ixekizumab (Experimental): Participants received Ixekizumab during the double-blind and extended treatment periods (i.e.,) starting dose of 160 milligrams (mg) Ixekizumab in the beginning week followed by 80 mg Ixekizumab once every four weeks (Q4W) by subcutaneous injection. No treatments were administered during the follow-up period.
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Participants received placebo every four weeks (Q4W) by subcutaneous (SC) injection during the double-blind period. During the extension period, they received starting dose of 160 milligrams (mg) Ixekizumab in the beginning week followed by 80 mg Ixekizumab once every four weeks (Q4W) by subcutaneous injection. No treatments were administered during follow-up period.
  Interventions: Drug: Ixekizumab; Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of ixekizumab in Chinese participants with radiographic axial spondyloarthritis (r-axSpA).

ELIGIBILITY:
Inclusion Criteria:

* Have an established diagnosis of radiographic axial spondyloarthritis (r-xSpA) with sacroiliitis defined radiographically according to the modified New York criteria.
* Participants have a history of back pain ≥3 months with age at onset <45 years.
* Biologic naïve or have had prior treatment with 1 tumor necrosis factor (TNF) inhibitor.
* Must have had an inadequate response to 2 or more NSAIDs at the therapeutic dose range for a total duration of at least 4 weeks OR have a history of intolerance to NSAIDs.
* Have a history of prior therapy for axSpa for at least 12 weeks prior to screening.

Exclusion Criteria:

* Have total ankylosis of the spine.
* Have recently received a live vaccine within 12 weeks or have had a vaccination with Bacillus Calmette-Guerin (BCG) within the past year.
* Have an ongoing or serious infection within the last 12 weeks.
* Have a compromised immune system.
* Have any other serious and/or uncontrolled diseases.
* Have either a current diagnosis or a recent history of malignant disease.
* Have had major surgery within 8 weeks of baseline, or will require surgery during the study.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- China (19):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - 1st Hospital affiliated to Medical College of Shantou Univer, Shantou, Guangzhou
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wu Han Tongji Hospital, Wuhan, Hubei
  - ZhuZhou Central Hospital, Zhuzhou, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - HuaShan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Beijing Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zhu X, Hu J, Liu D, Li J, Wu H, Sun L, Dai L, Tan C, Li Z, Xiao Z, Wang Y, Dong L, Yan Y, Li H, Zou H. Efficacy of Ixekizumab in Chinese Patients with Radiographic-Axial Spondyloarthritis by Baseline Inflammation Status on Magnetic Resonance Imaging. Rheumatol Ther. 2026 Jan 6. doi: 10.1007/s40744-025-00819-w. Online ahead of print. PMID 41495585
- [Derived] Kong N, Hu J, Liu D, Li J, Wu H, Sun L, Lie D, Tan C, Li Z, Xiao Z, Huang C, Xu J, Yan Y, Li H, Zou H. Efficacy of Ixekizumab in Chinese Patients with Radiographic Axial Spondyloarthritis by Baseline C-Reactive Protein Level. Rheumatol Ther. 2025 Aug;12(4):627-639. doi: 10.1007/s40744-025-00765-7. Epub 2025 May 9. PMID 40343690
- [Derived] Zhu X, Hu J, Liu D, Li J, Wu H, Sun L, Dai L, Tan C, Li Z, Xiao Z, Li X, Yan Y, Dou G, Sun Y, Zou H. Rapid and Sustained Effect of Ixekizumab on Patient Global, Spinal Pain, Stiffness, and Fatigue in Chinese Patients with Radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Aug;11(4):1011-1022. doi: 10.1007/s40744-024-00688-9. Epub 2024 Jun 21. PMID 38907104
- [Derived] Xue Y, Hu J, Liu D, Li J, Wu H, Tan C, Dai L, Sun L, Li Z, Xiao Z, Huang C, Yan Y, Ji F, Chen R, Zou H. Ixekizumab for Active Radiographic Axial Spondyloarthritis in Chinese Patients: 16- and 52-Week Results from a Phase III, Randomized, Double-Blind, Placebo-Controlled Study. BioDrugs. 2024 Jan;38(1):145-156. doi: 10.1007/s40259-023-00625-2. Epub 2023 Sep 22. PMID 37737952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to be conducted in three periods:
  * Double-Blind Treatment Period (Week 0 to Week 16)
  * Extended Treatment Period (Week 16 to Week 52)
  * Follow-up Period (at least 4 weeks and up to 12 weeks after the date of the participant's last visit)
Groups:
- Placebo: Participants received placebo every four weeks (Q4W) by subcutaneous (SC) injection.
- Ixekizumab 80mg Q4W: Participants received starting dose of 160 milligrams (mg) Ixekizumab at week 0 followed by 80mg Ixekizumab once every four weeks (Q4W) by subcutaneous injection.
- Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period: Participants from the "Placebo double-blind period" entered the extended treatment period where they received starting dose of 160 mg Ixekizumab at week 16 followed by 80 mg Ixekizumab Q4W by subcutaneous injection.
- Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period: Participants from the "Ixekizumab 80mg Q4W double-blind period" entered the extended treatment period where they continued receiving the same treatment.
- Placebo - Follow-up Period: Participants from the placebo arm entered the follow-up phase and were observed for safety. No treatments were administered.
- Ixekizumab 80mg Q4W - Follow-up Period: Participants from the Ixekizumab treated arms (Ixekizumab 80mg Q4W, Placebo/Ixekizumab 80mg Q4W, Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W arms) entered the follow-up phase and were observed for safety. No treatments were administered.
Period: Double-Blind Treatment Period
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period | Placebo - Follow-up Period | Ixekizumab 80mg Q4W - Follow-up Period
Started | 73 | 74 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 73 | 74 | 0 | 0 | 0 | 0
Completed | 71 | 74 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0
Period: Extended Treatment Period
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period | Placebo - Follow-up Period | Ixekizumab 80mg Q4W - Follow-up Period
Started | 0 (Double-blind treatment period arm.) | 0 (Double-blind treatment period arm.) | 70 (Participants from the double-blind treatment period who entered the extended treatment period.) | 72 (Participants from the double-blind treatment period who entered the extended treatment period.) | 0 | 0
Completed | 0 | 0 | 69 | 64 | 0 | 0
Not Completed | 0 | 0 | 1 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period | Placebo - Follow-up Period | Ixekizumab 80mg Q4W - Follow-up Period
Started | 0 | 0 | 0 (Extended treatment period arm.) | 0 (Extended treatment period arm.) | 1 (Participants from the double-blind or the extended treatment periods who entered the follow-up period.) | 135 (Participants from the double-blind or the extended treatment periods who entered the follow-up period.)
Completed | 0 | 0 | 0 | 0 | 0 | 123
Not Completed | 0 | 0 | 0 | 0 | 1 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Covid-19 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Ixekizumab 80mg Q4W: Participants received starting dose of 160 milligrams (mg) Ixekizumab at week 0 followed by 80 mg Ixekizumab once every four weeks (Q4W) by subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (8.98) | 33.5 (8.89) | 33.9 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 65 | 64 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 73 | 74 | 147
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 73 | 74 | 147
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 73 | 74 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society 40 (ASAS40) Response in Biological Disease-modifying Antirheumatic Drug (bDMARD)-naïve Participants
Description: ASAS40 is defined as improvement from baseline of greater than or equal to (>=) 40 % and absolute improvement from baseline of at least 2 units (range of 0 to 10) in at least 3 of the following 4 domains without any worsening in the remaining domain.
  1. Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  2. Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  3. Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function.
  4. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 16
Population: All randomized participants from bDMARD-naïve who had data for ASAS40.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 64 | 66
Percentage of Participants | 7.8 | 40.9
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.64, 95% CI 2-sided [2.68 to 21.76]

2. Secondary Outcome: Percentage of Participants Achieving an ASAS40 Response
Description: as for outcome 1
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Percentage of Participants | 8.2 | 37.8
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.40, 95% CI 2-sided [2.42 to 16.90]

3. Secondary Outcome: Percentage of Participants Achieving an ASAS20 Response
Description: ASAS20 response is defined as a ≥20% improvement and an absolute improvement from baseline of ≥1 units (range 0 to 10) in ≥3 of 4 domains, and no worsening of ≥20% and ≥1 unit (range 0 to 10) in the remaining domain.
  1. Patient Global: How active was your spondylitis on average during the last week? score ranges 0 (not active) to 10 (very active).
  2. Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  3. Bath Ankylosing Spondylitis Functional Index (BASFI): Participant asked to rate the difficulty associated with 10 individual basic functional activities. Participant response was captured using Numeric Rating Scale (NRS) (range 0 to 10) with a higher score indicating worse function.
  4. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Participants received placebo every four weeks (Q4W) by subcutaneous (SC)injection.
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Percentage of Participants | 35.6 | 59.5
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.31 to 5.09]

4. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with CRP as acute phase reactant) are
  1. Total back pain
  2. Patient global
  3. Peripheral pain/swelling
  4. Duration of morning stiffness and
  5. CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher scores indicated higher disease activity. Least Square (LS) mean was determined by mixed-model repeated measures (MMRM) with treatment, baseline C-reactive protein (CRP) status, Tumor necrosis factor (TNF) inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for ASDAS.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Units on a scale | -0.19 (0.103) | -1.33 (0.100)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.14, 95% CI 2-sided [-1.38 to -0.90], Standard Error of Mean 0.120

5. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Response
Description: The BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to radiographic axial spondyloarthritis (rad-axSpA): 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10 (NRS). Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe AS symptom. LS mean was determined by MMRM with treatment, baseline CRP status, TNF inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for BASDAI.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Units on a scale | -0.90 (0.231) | -2.39 (0.226)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.49, 95% CI 2-sided [-2.04 to -0.94], Standard Error of Mean 0.280

6. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a participant-reported assessment that establishes a participant's functional baseline and subsequent response to treatment. The BASFI is composed with 10 questions to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of AS participants. Participants respond to each question using an NRS scale (range 0 to 10). The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 10, with a higher score indicating worse function. LS mean was determined by MMRM with treatment, baseline CRP status, TNF inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for BASFI.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Placebo: Participants received placebo every four weeks (Q4W) by subcutaneous (SC)injection during.
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Units on a scale | -0.49 (0.237) | -1.36 (0.230)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.002, Mixed Models Analysis; LS Mean Difference = -0.87, 95% CI 2-sided [-1.43 to -0.32], Standard Error of Mean 0.280

7. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score)
Description: MRI score of spine was assessed using SPARCC method. All 23 disco-vertebral units (DVU) of the spine (from C2 to S1) were scored for bone marrow edema. A single DVU has 18 scoring units, and each has score of 0 or 1, bringing the maximum total score to 414, the sum ranges from 0 to 414 with higher scores reflecting worse disease. Scoring was performed by central readers. LS mean was determined by ANCOVA with factors for treatment, baseline CRP status, TNF inhibitors experience, and baseline value.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for MRI of the Spine.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 70 | 72
Units on a scale | -0.93 (1.550) | -8.65 (1.507)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -7.72, 95% CI 2-sided [-10.85 to -4.60], Standard Error of Mean 1.580

8. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: SF-36 consists of 36 questions measuring 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health perceptions, mental health, social function, and vitality. The patient's responses are solicited using Likert scales that vary in length, with 3-6 response options per item. The SF-36 can be scored into the 8 health domains named above and two overall summary scores: physical component summary (PCS) and mental component summary (MCS) scores. The domain and summary scores range from 0 to 100; higher scores indicate better levels of function and/or better health. LS mean was determined by MMRM with factors for treatment, baseline CRP status, TNF inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for SF-36 PCS score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 72 | 74
Units on a scale | 1.23 (0.740) | 3.85 (0.716)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.001, Mixed Models Analysis; LS Mean Difference = 2.62, 95% CI 2-sided [1.07 to 4.17], Standard Error of Mean 0.785

9. Secondary Outcome: Change From Baseline in 36-Item SF-36 Mental Component Summary (MCS) Score
Description: as for outcome 8
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for SF-36 MCS score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 72 | 74
Units on a scale | -0.06 (1.027) | 0.45 (1.003)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.660, Mixed Models Analysis; LS Mean Difference = 0.51, 95% CI 2-sided [-1.77 to 2.79], Standard Error of Mean 1.152

10. Secondary Outcome: Change From Baseline in the Measure of High Sensitivity C-Reactive Protein (CRP)
Description: High sensitivity CRP is the measure of acute phase reactant. It was measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on disease activity. High sensitivity CRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation. LS mean was determined by MMRM with treatment, baseline CRP status, TNF inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for CRP.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
milligram per liter (mg/L) | 2.65 (1.349) | -10.10 (1.312)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.75, 95% CI 2-sided [-15.91 to -9.59], Standard Error of Mean 1.594

11. Secondary Outcome: Change From Baseline in Mobility on the Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: BASMI is a combined index comprising of 5 clinical measurements of spinal mobility in patients with radiographic axial spondyloarthritis (rad-axSpA).
  1. Lateral Spinal Flexion
  2. Tragus-to-wall distance
  3. Lumbar Flexion (modified Schober)
  4. Maximal intermalleolar distance and
  5. Cervical rotation. The BASMI linear result is the average of the 5 assessments and ranges from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their AS. LS mean was determined by MMRM with treatment, baseline CRP status, TNF inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for BASMI.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 70 | 72
Units on a scale | 0.06 (0.093) | -0.30 (0.090)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.36, 95% CI 2-sided [-0.57 to -0.15], Standard Error of Mean 0.106

12. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Description: The MASES is an index used to measure the severity of enthesitis. The MASES assesses 13 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include costochondral 1 (right/left), costochondral 7 (right/left), spinal iliaca anterior superior (right/left), crista iliaca (right/left), spina iliaca posterior (right/left), processus spinosus L5, and Achilles tendon proximal insertion (right/left). The MASES is the sum of all site scores (range 0 to 13); higher scores indicate more severe enthesitis. LS mean was determined by MMRM with treatment, baseline CRP status, TNF inhibitors experience, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for MASES.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 41 | 33
Units on a scale | -1.06 (0.349) | -1.77 (0.361)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p = 0.086, Mixed Models Analysis; LS Mean Difference = -0.72, 95% CI 2-sided [-1.54 to 0.10], Standard Error of Mean 0.413

13. Secondary Outcome: Change From Baseline in MRI Sacroiliac Joint(s) (SIJ) Spondyloarthritis Research Consortium of Canada (SPARCC) Score
Description: The SPARCC enthesitis is an index used to measure the severity of enthesitis. The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis. LS mean was determined by ANCOVA with factors for treatment, baseline CRP status, TNF inhibitors experience, and baseline value.
Time Frame: Baseline, Week 16
Population: All randomized participants who had baseline and post-baseline data for MRI Sacroiliac Joint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 70 | 72
units on a scale | -1.31 (1.021) | -6.98 (0.986)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -5.67, 95% CI 2-sided [-7.71 to -3.62], Standard Error of Mean 1.034

14. Secondary Outcome: Number of Participants With Anterior Uveitis
Description: Anterior uveitis is an inflammation of the middle layer of the eye. which includes the iris (colored part of the eye) and the adjacent tissue, known as the ciliary body.
Time Frame: Baseline through Week 16
Population: All randomized participants who had data for Anterior Uveitis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Participants | 0 | 0

15. Secondary Outcome: Change From Baseline in ASAS-Nonsteroidal Anti-Inflammatory Drug (NSAID) Score
Description: ASAS-NSAID score is used to present the NSAID intake by considering the type of NSAID, the total dose and the number of days taking NSAID during a period of interest (PI). For the NSAID equivalence scoring system, "no NSAID intake" was set to a score value of 0, and the reference dose of NSAID (150 mg/day diclofenac) was set to a score value of 100. The Daily diclofenac-equivalent dose score was derived by converting each daily dose of NSAID to a percentage dose equivalent of 150 mg diclofenac. ASAS-NSAID score = (equivalent NSAID score) x (days of intake during PI) x (days per week)/(PI in days). The total score range is from 0 to 100, higher the score greater the NSAID intake and 0 represents no intake at all. A negative change from baseline indicates less NSAID consumption.
Time Frame: Baseline, Week 52
Population: Participants from extended treatment period who had NSAID intake at baseline and week 52.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period
Number analyzed (Participants) | 58 | 63
Units on a scale | -30.71 (46.481) | -26.13 (41.384)

16. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: A treatment emergent - antidrug antibody (TE-ADA) positive participant is defined as: a) a participant with a >= 4-fold increase over a positive baseline antibody titer; or b) for a negative baseline titer, a participant with an increase from the baseline to a level of >= 1:10. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Week 16
Population: All randomized participants who had data for Anti-Ixekizumab Antibodies.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 73 | 74
Percentage of participants | 4.1 | 13.5

17. Secondary Outcome: Pharmacokinetics (PK): Trough Ixekizumab Concentration at Steady State (Ctrough ss)
Description: Pharmacokinetics (PK): Steady-state trough serum concentration of Ixekizumab at week 16.
Time Frame: Week 16
Population: All randomized participants who received at least one dose and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliters (µg/mL)
Arm/Group | Ixekizumab 80mg Q4W
Number analyzed (Participants) | 74
microgram per milliliters (µg/mL) | 3.89 (52)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 64 Weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Placebo - Follow-up Period: Participants from the placebo arm who entered the follow-up phase were observed for safety. No treatments were administered.
- Ixekizumab 80mg Q4W - Follow-up Period: Ixekizumab treated participants (Ixekizumab 80mg Q4W, Placebo/Ixekizumab 80mg Q4W, Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W arms) who entered the follow-up phase were observed for safety. No treatments were administered.
Arm/Group | Placebo | Ixekizumab 80mg Q4W | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period | Placebo - Follow-up Period | Ixekizumab 80mg Q4W - Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/74 | 0/70 | 0/72 | 0/1 | 0/135
Serious Adverse Events (participants affected / at risk) | 1/73 | 2/74 | 6/70 | 4/72 | 0/1 | 1/135
Other Adverse Events (participants affected / at risk) | 17/73 | 31/74 | 43/70 | 41/72 | 0/1 | 11/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=73) | Ixekizumab 80mg Q4W (N=74) | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period (N=70) | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period (N=72) | Placebo - Follow-up Period (N=1) | Ixekizumab 80mg Q4W - Follow-up Period (N=135)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Male genital tract tuberculosis (Infections and infestations) | 0/65 (0) | 0/64 (0) | 1/62 (1) | 0/62 (0) | 0 (0) | 0/119 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Auricular haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign connective tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=73) | Ixekizumab 80mg Q4W (N=74) | Placebo/Ixekizumab 80mg Q4W - Extended Treatment Period (N=70) | Ixekizumab 80mg Q4W/Ixekizumab 80mg Q4W - Extended Treatment Period (N=72) | Placebo - Follow-up Period (N=1) | Ixekizumab 80mg Q4W - Follow-up Period (N=135)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 6 (7) | 3 (6) | 2 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 5 (7) | 20 (64) | 25 (81) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (13) | 9 (12) | 19 (21) | 16 (22) | 0 (0) | 5 (5)
Vaginal infection (Infections and infestations) | 0/8 (0) | 0/10 (0) | 1/8 (1) | 0/10 (0) | 0 (0) | 0/16 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (4) | 4 (4) | 3 (3) | 0 (0) | 2 (2)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4) | 6 (7) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 6 (7) | 7 (8) | 4 (4) | 0 (0) | 4 (4)
Pelvic fluid collection (Reproductive system and breast disorders) | 0/8 (0) | 0/10 (0) | 1/8 (1) | 0/10 (0) | 0 (0) | 0/16 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT04285229/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT04285229/SAP_001.pdf